CLINICAL TRIAL: NCT06168305
Title: Safety and Effectiveness of GENOSS® DES (Sirolimus-eluting Coronary Stent System) in Patients With Multivessel Coronary Artery Disease (MVCAD): A Multicenter, Prospective, Observational Study
Brief Title: Safety and Effectiveness of GENOSS® DES in Patients With Multivessel Coronary Artery Disease
Acronym: GENOSS-MV
Status: Enrolling by invitation | Type: Observational
Sponsor: Genoss Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023GR0399
Record Dates: First submitted 2023-11-28; First posted 2023-12-13 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Percutaneous Coronary Intervention; Multivessel Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GENOSS® DES Sirolimus Eluting Coronary Stent System / B03300.20, class [4]: Patients with multivessel coronary artery disease (MVCAD) who underwent percutaneous coronary intervention using GENOSS® DES
  Interventions: Device: GENOSS® DES Sirolimus Eluting Coronary Stent System

INTERVENTIONS:
Device: GENOSS® DES Sirolimus Eluting Coronary Stent System — The GENOSS® DES is L-605 cobalt chromium (CoCr) platform with a strut thickness of 70µm Sirolimus drug with concentration of 1.15µg/mm2 Abluminal biodegradable PLA and PLGA polymers.

SUMMARY:
The investigators intend to establish a multicenter prospective observational study by enrolling and tracking patients with multivessel coronary artery disease (MVCAD) using Genoss DES, a device manufactured with pure domestic technology. The study aims to evaluate the efficacy and safety of Genoss DES in MVCAD patients.

DETAILED DESCRIPTION:
This study is a sponsor-driven clinical trial (SIT) that aims to enroll patients who have undergone treatment for multivessel coronary artery disease using Genoss stents. The study involves collecting data on the clinical and surgical processes of patients and tracking the occurrence of clinical events.

This prospective, multicenter observational study registers patients with acute coronary artery disease who have been treated with GENOSS stents at a total of 8 institutions.

As it is an observational study, the number of subjects is not separately calculated, but the plan is to recruit a total of 1,000 participants during the study registration period.

ELIGIBILITY:
<Inclusion Criteria>

* Adults over 19 years of age
* Subjects with multivessel coronary artery disease (MVCAD) (However, subject registration is possible even if the treatment area is restenosis or recurrent lesion, including new lesions)
* Subjects who underwent percutaneous coronary intervention (PCI) with GENOSS® DES
* Research subjects who agree to the research protocol and clinical follow-up plan, voluntarily decide to participate in this clinical study, and give written consent in the informed consent form.

(However, in the case of foreigners, only those who can speak Korean fluently and understand Korean documents such as the consent form are included.)

<Exclusion Criteria>

* Test subjects with known hypersensitivity or contraindications to the following drugs or substances: heparin, aspirin, clopidogrel, sirolimus, contrast medium (however, even subjects with hypersensitivity to contrast medium can be controlled by steroids and pheniramine) In this case, registration is possible, but if there is known anaphylaxis, it is excluded)
* When balloon angioplasty is performed on a stenotic area, the balloon cannot be expanded.
* Those whose remaining life expectancy is less than 1 year
* Expecting to become pregnant, pregnant or lactating woman
* The patient was admitted to the hospital due to cardiogenic shock and was predicted to have a low chance of survival based on medical judgment.

Subject

* If the researcher determines that the product is not suitable for this clinical study or may increase the risks associated with participation in the study.
* Foreigners who cannot speak Korean fluently and have difficulty understanding Korean documents

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with multivessel coronary artery disease (MVCAD) who underwent percutaneous coronary intervention using GENOSS® DES
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | at 12 months after the procedure
  The composite end point of cardiac death, TV-MI (target vessel-MI), and TLR (target lesion revascularization)

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) | at 12 months after the procedure
  The composite end point of death, myocardial infarction, target lesion revascularization
Cardiac death | at 12 months after the procedure
Non-cardiac death | at 12 months after the procedure
TV-MI (target vessel-myocardial infarction) | at 12 months after the procedure
Non-target vessel myocardial infarction | at 12 months after the procedure
ID-TVR (ischemia-driven target vessel revascularization) | at 12 months after the procedure
Non-ischemia driven target vessel revascularization | at 12 months after the procedure
Incidence rate of acute stent thrombosis within 24 hours, subacute stent thrombosis within 30 days, and late stent thrombosis at 1 year | within 24 hours, 30 days, 1 year
  Acute (within 24 hours), subacute (within 30 days), late (within 1 year)
Device success | during the procedure
  The clinical device is successfully delivered to the target lesion, inflated normally, and recovered intact.
Procedure success | during the hospitalization period (up to 3 days)
  When the final residual lesion stenosis is less than 50% using any surgical method, and there is no post-procedural death, myocardial infarction, or revascularization during the hospitalization period.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University GURO Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No